CLINICAL TRIAL: NCT00358839
Title: Calcitonin Gene Related Peptide-Induced Headache in Patients With Familial Hemiplegic Migraine Type 1 and 2.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Collaborators: EUROHEAD (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: FHM-CGRP
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2006-11-10 (Estimated); Status verified 2006-11

CONDITIONS: Familial Hemiplegic Migraine
Keywords: Familial hemiplegic migraine type 1 and 2; CGRP; middle cerebral artery; superficial temporal artery; headache; genotype; Healthy Volunteers
MeSH Terms: conditions — Migraine with Aura; Hemiplegic migraine, familial type 1; Headache

INTERVENTIONS:
Drug: CGRP

SUMMARY:
The aim of the present study is to explore functional consequences of migraine gene mutations on their responses to Calcitonin Gene Related Peptide (CGRP)infusion.

DETAILED DESCRIPTION:
Calcitonin Gene Related Peptide (CGRP) induces migraine attacks indistinguishable from spontaneous attacks in approximately 50% of migraine sufferers. Treatment of spontaneous migraine attacks with an antagonist to CGRP is effective in many patients. These data show that CGRP is involved in both initiation and maintenance of migraine attack.

The consequence of migraine gene mutations on relevant migraine pathways has never been tested. The aim of the present study is to explore functional consequences of migraine gene mutations on their responses to CGRP infusion. The project will improve our understanding of the neurobiology of migraine and stimulate development of new treatment targets.

ELIGIBILITY:
Inclusion Criteria:

Patients: Diagnosis of familial hemiplegic migraine (IHS-classification criteria) caused by mutations in the CACNA1A gene and the ATP1A2 gene.

Controls: Healthy volunteers

Exclusion Criteria:

Controls: No primary headache in their own history 2) Patients and controls:

* A history of cerebrovascular disease and other CNS- disease
* A history of serious somatic and mental disease
* A history suggesting ischaemic heart disease
* A history of hypo- or hypertension
* Daily intake of medication apart from oral contraceptives
* Abuse of alcohol or medicine (opioid analgesics).
* Pregnant or breastfeeding women.

On the study day:

* No intake of a simple analgesic in the previous 48 hours
* No headache in the previous 48 hours

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2006-07; Study Completion 2006-10

PRIMARY OUTCOMES:
headache and associated symptoms
blood flow velocity of the middle cerebral artery
diameter of the superficial temporal artery

SECONDARY OUTCOMES:
MAP
HR

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Møller Hansen, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup, Copenhagen, Denmark